CLINICAL TRIAL: NCT01061528
Title: Distress Tolerance Treatment for Smoking Cessation
Brief Title: Coping Skills Treatment for Smoking Cessation
Acronym: Project-WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHI0906-002; R01DA017332 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Dependence
Keywords: cigarette smoking; smoking cessation; nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New Smoking Cessation Counseling (Experimental): * One 60-minute individual session
  * Seven 2-hour group sessions
  * Two individual brief telephone contacts over an eight-week period.
  * Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Interventions: Drug: Transdermal Nicotine
- Standard Smoking Cessation Counseling (Active Comparator): * One 60-minute individual session
  * Seven 2-hour group sessions
  * Two individual brief telephone contacts over an eight-week period.
  * Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Interventions: Drug: Transdermal Nicotine

INTERVENTIONS:
Drug: Transdermal Nicotine — Participants will use the full strength 21mg. patch for 4 weeks, will taper to the 14 mg. patch for the next 2 weeks, and then to the 7 mg. patch for the remaining 2 weeks of treatment.
  Other Names: Nicoderm CQ

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of a new type of exposure- and acceptance-based smoking cessation treatment vs. standard behavioral smoking cessation treatment, in conjunction with the use of the transdermal nicotine patch. In both treatments, participants will receive one 60-minute individual session, seven 2-hour group sessions and two individual brief telephone contacts over an eight-week period. Both treatments include 8 weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue after the treatment sessions have ended. Participants will provide follow-up data with regard to their smoking status through a one-year follow-up period.

DETAILED DESCRIPTION:
1. 18-65 years of age,
2. a regular smoker for at least one year,
3. currently smoking 10 or more cigarettes per day,
4. report motivation to quit smoking in the next month.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* regular smoker for at least one year
* currently smoking 10 or more cigarettes per day

Exclusion Criteria:

* Current Axis I disorder
* Psychoactive substance abuse or dependence (excluding nicotine dependence) within past year
* Current suicidal risk
* Pregnancy or breast feeding
* Use of nicotine replacement products or bupropion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Brown, PhD, Principal Investigator — Butler Hospital/Brown Medical School
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Distress Tolerance Cessation Counseling; Standard Smoking Cessation Counseling: One 60-minute individual session Seven 2-hour group sessions Two individual brief telephone contacts over an eight-week period. Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Transdermal Nicotine: Participants will use the full strength 21mg. patch for 4 weeks, will taper to the 14 mg. patch for the next 2 weeks, and then to the 7 mg. patch for the remaining 2 weeks of treatment.
Period: Overall Study
Arm/Group | Distress Tolerance Cessation Counseling | Standard Smoking Cessation Counseling
Started | 62 | 54
Completed | 59 | 52
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: Analysis population is not different from the assignment in Participant Flow.
Groups:
- New Smoking Cessation Counseling; Standard Smoking Cessation Counseling: * One 60-minute individual session
  * Seven 2-hour group sessions
  * Two individual brief telephone contacts over an eight-week period.
  * Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Transdermal Nicotine: Participants will use the full strength 21mg. patch for 4 weeks, will taper to the 14 mg. patch for the next 2 weeks, and then to the 7 mg. patch for the remaining 2 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | New Smoking Cessation Counseling | Standard Smoking Cessation Counseling | Total
Number analyzed (Participants) | 62 | 54 | 116
Age, Categorical [Count of Participants; unit: Participants] — The measure is a count of the number of participants enrolled in the study at baseline.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 62 | 54 | 116
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.97 (11.45) | 47.31 (10.98) | 46.06 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 36 | 32 | 68
Region of Enrollment [Number; unit: participants]
  United States | 62 | 54 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemically Verified Smoking Abstinence
Description: 1. Carbon monoxide of expired air
  2. Salivary cotinine level of saliva
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Tolerance Cessation Counseling | Standard Smoking Cessation Counseling
Number analyzed (Participants) | 62 | 54
Participants | 11 | 12

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Description: Definition of adverse event and/or serious adverse event does not differ from clinicaltrials.gov definitions. There were no adverse events reported during the course of the study.
Arm/Group | Distress Tolerance Cessation Counseling | Standard Smoking Cessation Counseling
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/54
Other Adverse Events (participants affected / at risk) | 0/62 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No